CLINICAL TRIAL: NCT04332224
Title: Efficacy of Blanketrol III and Arctic Sun in Cooling Non-shivering Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS23118 (B2019:076)
Record Dates: First submitted 2020-03-26; First posted 2020-04-02 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2021-03

CONDITIONS: Body Temperature Changes
Keywords: brain cooling; medical body cooling devices; Brain protection; hypoxia
MeSH Terms: conditions — Body Temperature Changes; Hypoxia

STUDY DESIGN:
Intervention Model Description: Repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-shivering cooling group (Experimental): Cooling devices
  Interventions: Device: Blanketrol cooling device and water-perfused blankets; Device: Blanketrol and Kool Kit; Device: Arctic Sun

INTERVENTIONS:
Device: Blanketrol cooling device and water-perfused blankets — Blanketrol and water-perfused blankets
Device: Blanketrol and Kool Kit — Blanketrol cooling device with water-perfused vest, hood and lower body blanket
Device: Arctic Sun — Arctic Sun cooling device with gel cooling pads

SUMMARY:
This study compares three medical cooling devices for effectiveness of cooling the core of non-shivering subjects. This relates to common protocols to cool patients experiencing myocardial infarctions or stokes.

DETAILED DESCRIPTION:
Body core and brain cooling by 1-3°C has been used as an adjunct in treatment of stroke and myocardial infarction (MI) patients. Body surface cooling is simple and non-invasive however this process is difficult to implement effectively because skin cooling stimulates shivering heat production, a defense mechanism that protects the body core from cooling. It is sometimes necessary to pharmacologically inhibit shivering in order to cool the body from surface cooling strategies such as application of cold packs or cold water-perfused blankets or pads.

Two commercial cooling units that are currently used are: 1) the Blanketrol III with standard Gel Pad (Gentherm Inc.); and 2) the Arctic Sun with hydrogel coated pads (Arctic Sun). A new cooling attachment system has been developed for the Blanketrol III. The new Kool Kit includes a head wrap, and a vest and lower body blanket. The effectiveness of the Kool Kit has not been quantified or compared to the current two systems mentioned above.

Since shivering heat production attenuates core cooling, it must be eliminated in clinical or research settings where core cooling effectiveness is the main dependent variable. Previous studies from this laboratory (Laboratory for Exercise and Environmental Medicine) have used a human model for severe hypothermia which meperidine (Demerol) is infused to inhibit shivering. Under these conditions the primary core cooling capacity of a cooling system can be determined.

The investigators intend to evaluate the Tco cooling rate, in hospital treatment conditions, [ambient temperature (Ta) = 22ºC] during surface cooling of non-shivering subjects with either: 1) Blanketrol with Gel Pads; 2) Blanketrol with Kool Kit; or 3) an Arctic Sun cooling system.

The purpose is to compare the core cooling rates induced by three commercial surface cooling devices in non-shivering subjects. Because of the increased total surface area of the cooling pads and blankets, the investigators hypothesize that the Blanketrol with Kool Kit will have a greater rate of core cooling than the other two cooling systems tested.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, who answer "No" to all the questions on a Get Active Questionnaire (GAQ) and the "Medical Screening Questionnaire for Hypothermia Study'.
* Participants will also be interviewed to determine that they are free of any cardio- respiratory disease, Raynaud's Syndrome, or any other conditions that can be aggravated by cold exposure.
* Also, the study will include women of child bearing potential willing to use highly effective birth control during the trial. All women of child bearing potential will complete the "Research participant information for female subjects" and undergo a pregnancy test at screening.

Exclusion Criteria:

* Anyone who gives a positive answer to any question in the GAQ or Medical Screening Questionnaire for Hypothermia Study, or who has any cardio-respiratory disease, renal dysfunction, Raynaud's Syndrome, past recreational drug use or any other conditions that can be aggravated by cold exposure will be excluded.
* Subjects contraindicated for meperidine administration or who have any of the conditions listed below will also be excluded from the study.
* hypersensitivity to meperidine or any ingredients in the formulation
* known or suspected mechanical GI obstruction or any diseases/conditions that affect bowel transit
* suspected surgical abdomen (i.e. acute appendicitis or pancreatitis)
* severe CNS depression, head injury, increased cerebrospinal or intracranial pressure
* convulsive disorder, delirium tremens
* hypothyroidism
* prostatic hypertrophy or urethral stricture
* sickle cell anemia
* Addison's disease
* Pheochromocitoma
* Known sensitivity or intolerance to the drug metoclopramide
* Use of medications that might interact negatively with meperidine. Examples should include MAO inhibitors at the time of screening or within 14 days of screening; CNS depressants; phenytoin; cimetidine; ritonavir; aclyclovir; skeletal muscle relaxants.
* pregnant women, breastfeeding women, and women planning on becoming pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Esophageal temperature cooling rate | 120 minutes
  Rate at which esophageal temperature decreases
Skin heat exchange | 120 minutes
  Body surface heat flux

CONTACTS AND LOCATIONS:
Locations (1):
- 211 Max Bell Centre, University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Leclerc C, Talebian Nia M, Giesbrecht GG. Heat Transfer Capabilities of Surface Cooling Systems for Inducing Therapeutic Hypothermia. Ther Hypothermia Temp Manag. 2023 Sep;13(3):149-158. doi: 10.1089/ther.2023.0003. Epub 2023 Jun 5. PMID 37276032